CLINICAL TRIAL: NCT07365462
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, and Tolerability of NBI-1065890 in Adult Participants With Tardive Dyskinesia
Brief Title: Efficacy, Safety, and Tolerability of NBI-1065890 Versus Placebo in Adults With Tardive Dyskinesia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-1065890-TD2033; 2025-524104-30-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-22; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-09

CONDITIONS: Tardive Dyskinesia
Keywords: Tardive Dyskinesia; NBI-1065890
MeSH Terms: conditions — Tardive Dyskinesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NBI-1065890 (Experimental): Participants will receive NBI-1065890.
  Interventions: Drug: NBI-1065890
- Placebo (Placebo Comparator): Participants will receive placebo matching NBI-1065890.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBI-1065890 — Oral administration
  Arms: NBI-1065890
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of NBI-1065890 compared with placebo for the treatment of tardive dyskinesia (TD) in adult participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Medically confirmed diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or major depressive disorder (MDD) as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) for at least 3 months prior to screening.
* Medically confirmed diagnosis of neuroleptic-induced TD as defined in the DSM-5 for at least 3 months prior to screening.
* Moderate or severe TD (AIMS Item 8, severity of abnormal movement overall) as assessed by a blinded, external AIMS video reviewer using a video recording of the participant's AIMS assessment administered at the clinical site by a blinded, certified site AIMS rater. The AIMS dyskinesia total score (sum of Items 1 to 7) must be ≥6 as assessed by the blinded, external AIMS video reviewer.

Key Exclusion Criteria:

* Comorbid parkinsonism (drug-induced or otherwise) or more than a minimal level of extrapyramidal signs/symptoms, as documented by a score on the Modified Simpson-Angus Scale (mSAS) (excluding Items 8 and 10) >6 at screening or Day -1 (baseline) or a score >3 in any one item (excluding Items 8 and 10).
* Barnes Akathisia Rating Scale (BARS) global clinical assessment score ≥2 at screening or Day -1.
* Brief Psychiatric Rating Scale (BPRS) total score ≥50 at screening or Day -1.
* Hospitalized for schizophrenia, schizoaffective disorder, bipolar disorder, or MDD within 6 months of screening.
* Participant has an unstable medical condition or unstable chronic disease.
* Any known history of neuroleptic malignant syndrome (NMS).

Note: Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Abnormal Involuntary Movement Scale (AIMS) Dyskinesia Total Score at Week 8 Based on the Blinded Central AIMS Video Raters' Assessment | Baseline and Week 8

SECONDARY OUTCOMES:
Percentage of Participants Who Are a Clinical Global Impression - Improvement (CGI-I) Responder 1 at Week 8 | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences